CLINICAL TRIAL: NCT06559241
Title: Safety and Efficacy of Remote Ischemic Conditioning for Acute Ischemic Stroke Treated With Mechanical Thrombectomy (RECAST-MT): A Multicenter, Randomized, Controlled, Open-label, Blinded Endpoint Trial
Brief Title: Remote Ischemic Conditioning for Acute Ischemic Stroke Treated With Mechanical Thrombectomy（RECAST-MT）
Acronym: RECAST-MT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECAST-MT
Record Dates: First submitted 2024-08-04; First posted 2024-08-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke; Anterior Circulation Brain Infarction
Keywords: Endovascular thrombectomy; Cerebroprotection; Remote ischemic conditioning
MeSH Terms: conditions — Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Patients in the control group will receive endovascular thrombectomy and the best medical management according to the guidelines.
  Interventions: Procedure: Endovascular thrombectomy; Drug: Best medical management
- 14-day treatment group (Experimental): Patients in the 14-day treatment group will receive endovascular thrombectomy and the best medical management according to the guidelines. In addition, this group will receive remote ischemic conditioning once pre-thrombectomy and twice daily for 14 days post-thrombectomy.
  Interventions: Device: 14-day remote ischemic conditioning; Procedure: Endovascular thrombectomy; Drug: Best medical management
- 30-day treatment group (Experimental): Patients in the 30-day treatment group will receive endovascular thrombectomy and the best medical management according to the guidelines. In addition, this group will receive remote ischemic conditioning once pre-thrombectomy and twice daily for 30 days post-thrombectomy.
  Interventions: Device: 30-day remote ischemic conditioning; Procedure: Endovascular thrombectomy; Drug: Best medical management

INTERVENTIONS:
Device: 14-day remote ischemic conditioning — RIC is a noninvasive therapy performed by an electric auto-control device with a cuff placed on the upper arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of the cuff on the upper arm. The procedure will be performed once before endovascular thrombectomy and twice daily for 14 days post-thrombectomy.
  Other Names: 14-day RIC
  Arms: 14-day treatment group
Device: 30-day remote ischemic conditioning — RIC is a noninvasive therapy performed by an electric auto-control device with a cuff placed on the upper arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of the cuff on the upper arm. The procedure will be performed once before endovascular thrombectomy and twice daily for 30 days post-thrombectomy.
  Other Names: 30-day RIC
  Arms: 30-day treatment group
Procedure: Endovascular thrombectomy — Endovascular thrombectomy procedures are performed according to the guidelines to recanalize the occluded large vessel safely.
  Other Names: EVT
Drug: Best medical management — Best medical management is prescribed at the discretion of the treating physicians according to the guidelines.

SUMMARY:
For patients with acute ischemic stroke caused by large vessel occlusion, endovascular thrombectomy has been demonstrated to be the most effective therapy, as approximately 90% of the occluded vessels can be recanalized. However, less than 50% of patients could achieve functional independence, and over 15% died 90 days after stroke. Although the mismatch of successful recanalization with poor prognosis can be attributed to many factors, the infarct core formed during thrombectomy and reperfusion injury after thrombectomy may be among the most important and effective neuroprotective strategies urgently needed.

Remote ischemic conditioning (RIC) is a noninvasive strategy in which one or more cycles of brief and transient limb ischemia confer protection against prolonged and severe ischemia in distant organs. In the transient focal cerebral ischemia-reperfusion model, the application of remote ischemic conditioning before reperfusion or both before and after reperfusion reduces reperfusion injuries and the final infarct size. Because patients with acute ischemic stroke who are treated with endovascular thrombectomy can achieve a high rate of recanalization after focal ischemia, this patient population is akin to the model of transient focal cerebral ischemia-reperfusion. Furthermore, a pilot study has determined the safety and feasibility of remote ischemic conditioning in patients undergoing endovascular thrombectomy. However, whether remote ischemic conditioning could provide clinical benefits to patients with acute ischemic stroke who are treated with endovascular thrombectomy urgently needs investigations.

This study aims to investigate the safety and efficacy of remote ischemic conditioning in improving functional outcomes of patients with acute ischemic stroke treated with endovascular thrombectomy and explore the effect of treatment duration on the treatment outcome of remote ischemic conditioning.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years；
2. Acute ischemic stroke due to large vessel occlusion in the anterior circulation that is not suitable for intravenous thrombolytic therapy, or has contraindications to intravenous thrombolytic therapy, or treated with intravenous thrombolytic therapy without recanalization;
3. Large vessel occlusion confirmed by computed tomography angiography (CTA) or magnetic resonance angiography (MRA), including the occlusion of the intracranial segment of the internal carotid artery (ICA) and M1 segment of the middle cerebral artery (MCA), is the cause of symptoms, and mechanical thrombectomy is planned within 24 hours from the time last known well;
4. Baseline score of the National Institutes of Health Stroke Scale (NIHSS) ≥ 6 points;
5. Patients or family members signed a written informed consent form.

Exclusion Criteria:

1. Imaging examination revealed the presence of multiple vascular supply areas of cerebral infarction (such as the simultaneous presence of infarction in both anterior and posterior circulation);
2. Absence of femoral artery pulsation, extremely difficult intravascular access, or extremely tortuous large vessels, which are expected to result in the inability to undergo timely endovascular treatment;
3. Difficult-to-control hypertension: continuous monitoring upon admission shows systolic blood pressure ≥180mmHg, or diastolic blood pressure ≥100mmHg;
4. Coma or lethargy patients (consciousness level score ≥2 in NIHSS);
5. Unable to obtain an accurate baseline NIHSS score;
6. Pre-stroke modified Rankin Scale (mRS) score >1;
7. Baseline ASPECTS score ≤5;
8. Presence of bleeding tendency, deficiency of coagulation factors, or oral anticoagulant therapy with INR > 3.0;
9. Baseline blood glucose <2.7mmol/L or >22.2mmol/L;
10. Baseline platelet count < 30*10^9/L;
11. Severe known renal impairment defined as requiring dialysis (hemodialysis or peritoneal dialysis), or if known creatinine clearance rate <30mL/min;
12. Cranial CT or MRI shows intracranial hemorrhage;
13. Cranial CT or MRI shows midline deviation and significant occupying effect;
14. Clinical history, previous imaging examinations, or clinical judgment suggesting intracranial tumors, arteriovenous malformations, or intracranial arterial dissection;
15. History of head injury in the past 3 months;
16. History of life-threatening allergy to contrast agents, nickel, titanium metal, or their alloys;
17. Pregnancy, if women of childbearing age have a positive urinary or serum β-human chorionic gonadotropin (β-hCG) test or are breastfeeding；
18. The life expectancy of patients is less than 6 months, and they cannot be evaluated within 3 months;
19. Limb deformity, soft tissue injury, or other conditions that affect the implementation of distant ischemia adaptation therapy;
20. Participating in other ongoing clinical trials;
21. Other conditions that the investigators believe are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2105 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving a modified Rankin Scale (mRS) score of 0-2 at 90 days. | 90 days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Two dichotomous mRS scores at 90 days (0-1 vs 2-6, 0-3 vs 4-6, 0-4 vs 5-6, 0-5 vs 6). | 90 days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating worse outcomes.
The ordinal distribution of mRS scores at 90 days. | 90 days after stroke.
  The mRS ranges from 0 to 6, with higher scores indicating worse outcomes.
The proportion of patients with early neurological improvement 24 hours after endovascular procedures. | 24 hours after endovascular procedures.
  The NIHSS ranges from 0 to 42, with higher scores indicating worse outcomes. Neurological improvement is defined as the NIHSS recovering to ≤2 points or decreasing by 8 points or much higher as compared with the baseline.
Changes in NIHSS score from baseline to day 14 or at discharge (whichever comes earlier). | 14 days or at discharge (whichever comes first)
  The NIHSS ranges from 0 to 42, with higher scores indicating worse outcomes.
Score of EQ-5D-5L at 90 days. | 90 days after stroke.
  EQ-5D-5L is a tool used to assess health status, including five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A higher score indicates a better health status, while a lower score indicates a poorer health status.
Cerebral infarct volume. | 72 hours after endovascular procedures.
  The infarction volume will be assessed on cranial CT or MRI imaging.
The change of infarct volume. | 72 hours after endovascular procedures.
  Infarct Expansion Ratio (IER, IER=infarct volume/baseline infarct volume). The infarction volume will be assessed on cranial CT or MRI imaging, and baseline infarct volume will be assessed on the CTP or baseline MRI imaging.
Incidence of intracranial hemorrhage. | Within 14 days after endovascular procedures.
  Intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging, according to the criteria of the ECASS III.
Incidence of Symptomatic Intracranial Hemorrhage | Within 14 days after endovascular procedures.
  Symptomatic intracranial hemorrhage is defined as the demonstration of hemorrhage within brain parenchyma on head imaging leading to an increase of at least 4 points in the NIHSS score, according to the criteria of the European Cooperative Acute Stroke Study III (ECASS III).
Incidence of neurological deterioration within 14 days. | Within 14 days after endovascular procedures.
  Neurological deterioration is defined as an increase of ≥4 points in NIHSS compared to before deterioration within 14 days.
Incidence of malignant infarction | 0-90 days
  Malignant infarction is defined as infarction involving more than half of the affected middle cerebral artery area, a significant mass effect requiring decompressive craniectomy, and/or directly leading to death with clinical signs of brain herniation.
All cause of death. | 0-90 days
  The incidence of death events at any time from randomization through day 90.
Incidence of Adverse Events/Serious Adverse Events | 0-90 days
  The incidence of other adverse events and serious adverse events at any time from randomization through day 90.

CONTACTS AND LOCATIONS:
Locations (56):
- China (56):
  - Suzhou Municipal Hospital of Anhui Province, Suzhou, Anhui
  - Taihe County People's Hospital, Taihe Chengguanzhen, Anhui
  - Tongling People's Hospital, Tongling, Anhui
  - Beijing Luhe Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Fangshan District First Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - South China Hospital Affiliated to Shenzhen University, Shenzhen, Guangdong
  - The Second Nanning People's Hospital, Nanning, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Army Medical University Noncommissioned Officer School Affiliated Hospital, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Hongda Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Xunxian People's Hospital, Hebi, Henan
  - Jiaozuo Coal Industry Group Co., Ltd. Central Hospital, Jiaozuo, Henan
  - Luoyang Yanshi People's Hospital, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Province People's Hospital, Zhengzhou, Henan
  - Xihua county people's hospital, Zhoukou, Henan
  - Huanggang Central hospital, Huanggang, Hubei
  - Huangshi central hospital, Huangshi, Hubei
  - Jingmen Central hospital, Jingmen, Hubei
  - Jingmen People's Hospital, Jingmen, Hubei
  - First People's Hospital of Tianmen, Tianmen, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third People's Hospital of Hubei Province, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - the First People's Hospital of Changde, Changde, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - the First People's Hospital of Chenzhou, Chenzhou, Hunan
  - The Central Hospital of Xiangtan, Xiangtan, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Anshan Changda Hospital, Anshan, Liaoning
  - Dalian Central Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Jinan Third People's Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Liaocheng Third People's Hospital, Liaocheng, Shandong
  - The People's Hospital of Gaotang, Liaocheng, Shandong
  - Feixian People's Hospital, Linyi, Shandong
  - Yeda Hospital, Yantai, Shandong
  - Mianyang third people's hospital, Mianyang, Sichuan
  - Ya 'an People's Hospital, Ya'an, Sichuan
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Yueqing People's Hospital, Yueqing, Zhejiang
  - Beijing Chao-Yang Hospital, Beijing
  - Aerospace Central Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Beijing Fengtai You'anmen Hospital, Beijing
  - Beijing Red Cross Emergency Medical Center, Beijing
  - Beijing Daxing District People's Hospital, Beijing
  - Chongqing University Fuling Hospital, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao W, Meng R, Ma C, Hou B, Jiao L, Zhu F, Wu W, Shi J, Duan Y, Zhang R, Zhang J, Sun Y, Zhang H, Ling F, Wang Y, Feng W, Ding Y, Ovbiagele B, Ji X. Safety and Efficacy of Remote Ischemic Preconditioning in Patients With Severe Carotid Artery Stenosis Before Carotid Artery Stenting: A Proof-of-Concept, Randomized Controlled Trial. Circulation. 2017 Apr 4;135(14):1325-1335. doi: 10.1161/CIRCULATIONAHA.116.024807. Epub 2017 Feb 7. PMID 28174194
- [Result] Zhao W, Wu C, Dornbos D 3rd, Li S, Song H, Wang Y, Ding Y, Ji X. Multiphase adjuvant neuroprotection: A novel paradigm for improving acute ischemic stroke outcomes. Brain Circ. 2020 Feb 18;6(1):11-18. doi: 10.4103/bc.bc_58_19. eCollection 2020 Jan-Mar. PMID 32166195
- [Result] An JQ, Cheng YW, Guo YC, Wei M, Gong MJ, Tang YL, Yuan XY, Song WF, Mu CY, Zhang AF, Saguner AM, Li GL, Luo GG. Safety and efficacy of remote ischemic postconditioning after thrombolysis in patients with stroke. Neurology. 2020 Dec 15;95(24):e3355-e3363. doi: 10.1212/WNL.0000000000010884. Epub 2020 Oct 7. PMID 33028663
- [Derived] Wang Y, Huang S, Liu L, Ji X, Zhao W, Li S; RECAST-MT investigators. Safety and Efficacy of Remote Ischaemic Conditioning for Acute Ischaemic Stroke Treated with Mechanical Thrombectomy (RECAST-MT): rationale and design. Stroke Vasc Neurol. 2025 Nov 25:svn-2025-004591. doi: 10.1136/svn-2025-004591. Online ahead of print. PMID 41290408